CLINICAL TRIAL: NCT02373787
Title: A 5 Year Clinical Investigation on Creos Xenoprotect
Acronym: CXP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T 186
Record Dates: First submitted 2014-10-20; First posted 2015-02-27 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Implant
Keywords: Resorbable; Collagen membrane; NobelReplace CC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- creos xenoprotect (Experimental): resorbable collagen membrane
  Interventions: Device: creos xenoprotect
- Bio-Gide (Active Comparator): Bio-Gide, resorbable collagen membrane
  Interventions: Device: Bio-Gide

INTERVENTIONS:
Device: creos xenoprotect — Implant placement with simultaneous bone augmentation
  Arms: creos xenoprotect
Device: Bio-Gide — resorbable collagen membrane
  Arms: Bio-Gide

SUMMARY:
A 5-year clinical investigation on creos xenoprotect

DETAILED DESCRIPTION:
Randomized, prospective, multi-center study evaluating creos xenoprotect versus Bio-Gide® for guided bone regeneration in dehiscence defects

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent from the subject.
* The subject shall be at least 18 years of age and has passed cessation of growth.
* The subject must be in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems.
* The patient is willing and able to comply with all study related procedures (such as exercising oral hygiene and attending all follow-up procedures).
* The subject requires a single unit implant restoration with guided bone regeneration in bony defects in the anterior and premolar areas of maxilla or mandible.
* If two or more site single unit implant restorations requiring bone augmentation are required, only one will be included in the study, the other site will be treated with standard of care.
* The subject shall be healthy and compliant with good oral hygiene.
* Full-mouth bleeding score (FMBS) lower than 25% [20].
* Full-mouth plaque score (FMPI) lower than 20% [21].
* The implant site is free from infection and extraction remnants.
* The subject shall have a favourable and stable occlusal relationship.
* Natural roots are adjacent to implant site.
* The subject is suitable for a 2-stage surgical procedure. Secondary inclusion criteria at time of surgery
* Sufficient bone volume at the implant site for placing a NobelReplace CC implant.
* Initial implant stability as assessed by hand testing.
* Defect size for guided bone regeneration:

Height ≥ 3 mm and ≤ 7 mm as assessed with a UNC15 periodontal probe.

Exclusion Criteria:

* Previous bone augmentation at the implant site.
* Extraction site less than 3 months after extraction.
* Soft tissue grafting at implant placement, soft tissue grafting is allowed only at re-entry.
* Health conditions, which do not permit the surgical treatment.
* Any disorders in the planned implant area such as previous tumours, chronic bone disease or previous irradiation
* Infections in the planned implantation site or adjacent tissue.
* Acute, untreated periodontitis in the planned implantation site or adjacent tissue.
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc).
* Alcohol or substance abuse as noted in subject records or in subject history.
* Heavy smoking (>10 cigarettes/day).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 8%.
* Severe bruxism or other destructive habits.
* Pregnant or lactating women at the time of collagen membrane insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01-28 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate bone regeneration through measurement of defect height | 6 months

SECONDARY OUTCOMES:
Adverse events (AEs) | 6 months

OTHER OUTCOMES:
Membrane Dehiscence | 6 months
success and survival rates of implants | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arrighi, PhD, Study Director — Nobel Biocare Services AG
Locations (1):
- Praxisklinik der Zahnheilkunde am Luisenhospital, Aachen, Germany